CLINICAL TRIAL: NCT06499649
Title: Randomized, Double-blind, Placebo-controlled Clinical Study to Assess the Adjuvant Role of Dietary Supplementation of Antibiotic-tolerant Probiotics in Standard Therapy for the Eradication of Helicobacter Pylori Infection.
Brief Title: Assessment of the Adjuvant Role of Dietary Supplementation of Antibiotic-tolerant Probiotics in Standard Therapy for the Eradication of Helicobacter Pylori Infection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IBSA Farmaceutici Italia Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IBSAHP_2024
Record Dates: First submitted 2024-07-08; First posted 2024-07-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Helicobacter Pylori Infection
Keywords: Probiotics; Dietary Supplementation; Eradication Therapy; Double-blinded

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): Patients under H. pylori eradication therapy and placebo as treatment
  Interventions: Dietary Supplement: Placebo
- Treated group (Experimental): Patients under H. pylori eradication therapy and probiotics as treatment
  Interventions: Dietary Supplement: IBSA Probiotics

INTERVENTIONS:
Dietary Supplement: IBSA Probiotics — Dietary supplement base on probiotic strains.
  Arms: Treated group
Dietary Supplement: Placebo — The placebo does not contain functional components, and the appearance is indistinguishable from the comparison product.
  Arms: Control group

SUMMARY:
Randomized, double-blind, placebo-controlled clinical study to assess the adjuvant role of dietary supplementation of antibiotic-tolerant probiotics, derived from Lactobacillus acidophilus and Bifidobacterium animalis, in standard therapy for the eradication of Helicobacter pylori infection.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled clinical study to assess the adjuvant role of dietary supplementation of antibiotic-tolerant probiotics, in standard therapy for the eradication of H. pylori infection.

The aim of this study is to evaluate the antibiotic adverse events decrease in subjects under the standard therapy for H. Pylori eradication using probiotics, compared to patients receiving the same antibiotic therapy with placebo.

This study is aimed to (naive) patients who have never received the eradication therapy.

The infection of H. Pylori will be analyzed using Urea Breath Test, esophagogastroduodenoscopy (EGDS), Histological and/or culture examination on biopsy samples.

The incidence and severity of the adverse events related to the eradication therapy will be assessed through the evaluation questionnaire EACTE (Eventi Avversi Correlati con la Terapia Eradicante) - Adverse Events correlated to Eradication Therapy.

The differences of Gastrointestinal Symptom Rating Scale (GSRS) score will be recorded to compare the two groups (patients under antibiotic therapy and probiotics/placebo treatment).

The study will involve 270 patients affected by H. pylori, with 1:1 ratio of probiotic/placebo treatment.

Each enrolled and randomized patient should take daily:

Probiotics or Placebo, depending on the treatment group assigned by randomization, (1 capsule twice a day before breakfast and dinner) for 10 days, before beginning eradication therapy. After the first 10 days of dietary supplementation with probiotics or placebo, the patient will be accompanied by dietary supplementation with eradication therapy (duration 10 days). At the end of the eradication therapy, the patient will continue feeding only probiotics or placebo for a further 4 weeks, with a dosage similar to that used before the beginning of the eradication therapy.

On the occasion of the T1 visit (after 20 days from T0 and to complete the eradication therapy), the following will be carried out:

* completion by the medical investigator of the EACTE questionnaire, on the basis of the patient's reports on any adverse events occurring during the study and related to eradication therapy, for the period between T0 and T1;
* check that the patient has taken the eradication therapy as indicated;
* registration of concurrent processing;
* recording of adverse events.

During the T2 visit (4 weeks after the end of the eradication therapy), the following will be carried out:

* urea breath test for the evaluation of HP eradication
* administration by the investigator of a questionnaire for the assessment of symptoms of functional dyspepsia, to be completed at T2 (GSRS questionnaire).
* recording of adverse events
* study conclusion Since this is a double-blind study, neither the doctor nor the patient will be aware of the nature of dietary supplementation (probiotic or placebo) assigned to the patient at T0.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of H. pylori infection by breath test and histological and/or cultural examination on biopsy (performed within 10 days prior to T0)
* Prescription of eradication therapy for HP
* Naïve patients (who have never had eradication therapy for H. pylori)
* Patients with symptoms of upper gastrointestinal tract
* Obtaining informed consent

Exclusion Criteria:

* Patients with history of previous eradication attempts
* Patients with known gastric disease (e.g. atrophic gastritis, gastric cancer)
* Patients with severe organ dysfunction (cirrhosis of the liver, severe renal or respiratory failure, dialysis)
* Women who are pregnant or breastfeeding
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
EACTE (Adverse Events Correlated to Eradication Therapy) incidence | T0 (basal) - T1 (20 ± 3 days after T0)
  Assessment of the incidence of "Adverse events related to eradication therapy" regardless of the degree of severity, in the group taking the dietary supplement with probiotic, compared to the group taking placebo. The adverse events related to eradication therapy are those described by the EACTE Assessment Questionnaire used

SECONDARY OUTCOMES:
EACTE severity | T0 (basal) - T2 (48 ± 3 days after T0)
  Assessment of the variation in severity of EACTE in the probiotic group compared to the placebo group.
Eradication rate of H. pylori | T2 (48 ± 3 days after T0)
  Percentage difference of eradication rate between placebo and treated groups
Severe EACTE | T0 (basal) - T1 (20 ± 3 days after T0)
  Difference between the percentage of subjects with at least one severe EACTE between the group taking probiotic treatment and the group taking placebo
GSRS (Gastrointestinal Symptom Rating Scale) score | T2 (48 ± 3 days after T0)
  Difference of GSRS score between placebo and treated groups.

OTHER OUTCOMES:
Safety Evaluation | T1 (20 ± 3 days after T0) and T2 (48 ± 3 days after T0)
  Adverse Events registration

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico S. Orsola - Malpighi - Università di Bologna, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided